CLINICAL TRIAL: NCT01176175
Title: Randomized, Controlled, Open-label, Parallel, Clinical Trial to Assess Pharmacokinetics and Endometrial Effect of an Injectable Formulation of Progesterone Microspheres in Doses of 50 mg, 100 mg, 200 mg and 300 mg, in Postmenopausal Women.
Brief Title: Progesterone Microspheres Pharmacokinetic - Pharmacodynamic (PK-PD) Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Productos Científicos S. A. de C. V. (Industry)
Responsible Party: Principal Investigator, Roberto Bernardo Escudero, Principal Investigator, Productos Científicos S. A. de C. V.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0908/I/PRO
Record Dates: First submitted 2010-08-04; First posted 2010-08-05 (Estimated); Last update posted 2011-10-13 (Estimated); Status verified 2011-10

CONDITIONS: Infertility
Keywords: Progesterone; Microspheres; postmenopausal; Luteal phase support
MeSH Terms: conditions — Infertility | interventions — Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 50 mg (Experimental): Progesterone microspheres injectable suspension 50 mg
  Interventions: Drug: Progesterone
- 100 mg (Experimental): Progesterone microspheres injectable suspension 100 mg
  Interventions: Drug: Progesterone
- 200 mg (Experimental): Progesterone microspheres injectable suspension 200 mg
  Interventions: Drug: Progesterone
- 300 mg (Experimental): Progesterone microspheres injectable suspension 300 mg
  Interventions: Drug: Progesterone

INTERVENTIONS:
Drug: Progesterone — Progesterone microspheres injectable suspension 50 mg, intramuscular weekly injection for a total of 7 doses.
  Arms: 50 mg
Drug: Progesterone — Progesterone microspheres injectable suspension 100 mg, intramuscular weekly injection for a total of 7 doses.
  Arms: 100 mg
Drug: Progesterone — Progesterone microspheres injectable suspension 200 mg, intramuscular weekly injection for a total of 7 doses.
  Arms: 200 mg
Drug: Progesterone — Progesterone microspheres injectable suspension 300 mg, intramuscular weekly injection for a total of 7 doses.
  Arms: 300 mg

SUMMARY:
Phase: I pharmacokinetic - pharmacodynamic (PK-PD) study. Main objective: To establish the minimum effective dose of progesterone microspheres suspension, which administered by weekly intramuscular injection, will be able to induce transformation from a proliferative endometrium to a secretory endometrium.

Study design: Randomized, controlled, open-label, parallel, dose-response clinical trial.

Sites: 1 Subjects: 48 postmenopausal women.

DETAILED DESCRIPTION:
Sites: 1 Phase: 1 Main objective:To establish the minimum effective dose of progesterone microspheres suspension, which administered by weekly intramuscular injection, will be able to induce transformation from a proliferative endometrium to a secretory endometrium.

Secondary objectives:

* To determine and compare the steady-state pharmacokinetic profile of investigational products.
* To evaluate safety profile of investigational products in the study subjects.
* To evaluate local tolerability of investigational products in the study subjects.

Study design:Randomized, controlled, open-label, parallel, dose-response clinical trial.

Investigational products:

* Progesterone microspheres intramuscular injectable suspension 50 mg
* Progesterone microspheres intramuscular injectable suspension 100 mg
* Progesterone microspheres intramuscular injectable suspension 200 mg
* Progesterone microspheres intramuscular injectable suspension 300 mg Study subjects: 48 healthy postmenopausal women, 45 - 60 years. Brief description: After written informed consent, 48 eligible women will receive pretreatment with oral estradiol valerate, then, 14 days later, those with adequate endometrial thickness evaluated through ultrasound will be randomized to study treatments (one IM injection each 7 days, for a total of 7 doses). 10 days after the first progesterone dose, an endometrial biopsy will be obtained. Blood samples will be obtained for pharmacokinetic study.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 45 to 60 years old
* Able to read and write
* Postmenopausal
* Body Mass Index equal or below 34.99 kg/m2
* Healthy
* Normal uterus
* Time availability

Exclusion Criteria:

* Hypersensitivity to progesterone or related compounds
* Hypersensitivity to estrogens
* Hysterectomy
* History or present hormone-dependent tumor
* History or present uterine cervix dysplasia
* Abnormal and clinically-significant laboratory test results
* Family history of breast cancer
* History of thromboembolic disease
* Non-controlled hypertension
* History of stroke
* History of cardiac valve surgery
* Renal failure
* Hepatic failure
* Non-controlled diabetes
* Severe gastrointestinal disease
* History of serious neurologic disease
* Reduced mobility
* Anemia
* Previous or concomitant hormonal therapy
* Previous or concomitant therapy with inhibitors or inductors of cytochrome

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2010-08; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Endometrial dating through histopathologic criteria. | 10 days
  Endometrial dating according Noyes criteria as a measure of efficacy. At the moment of the biopsy, study subjects would have received 25 days of estradiol valerate pretreatment and 10 days of progesterone (investigational product); thus simulating the 25th day of a menstrual cycle. Efficacy will be measured as number of biopsies that have histological date according to cronological date.

SECONDARY OUTCOMES:
Pharmacokinetics | 0 -60 days.
  Progesterone plasmatic concentrations and pharmacokinetic parameters.
Adverse events | 0 - 65 days
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability Pain Scores on a Visual Analog Scale

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Bernardo, MD MSc, Principal Investigator — Asociación Mexicana para la Investigación Clínica, A. C. (AMIC)
Locations (1):
- Asociación Mexicana para la Investigación Clínica, A. C. (AMIC), Pachuca, Hidalgo, Mexico